CLINICAL TRIAL: NCT01300611
Title: Phase I Evaluation of the Safety and Efficacy of TXA127 (Angiotensin 1-7) to Enhance Engraftment in Adults Undergoing Double Cord Blood Transplantation
Brief Title: TXA127 in Enhancement of Engraftment in Adult Double Cord Blood Transplantation
Acronym: USBTXA127CBT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Tarix Pharmaceuticals (Industry)
Collaborators: Constant Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TXA127-2010-001; NCT01302678 (obsolete NCT alias)
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Double Cord Blood Transplant; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Myelofibrosis; Acute Lymphoblastic Leukemia; Chronic Myelocytic Leukemia; Non Hodgkins Lymphoma; Hodgkins Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Double Cord Blood Transplantation; Neutrophil Engraftment; Platelet Engraftment; Immune Reconstitution; Mucositis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Mucositis | interventions — angiotensin I (1-7)

ARMS (2):
- TXA127 300 mcg/kg/day (Experimental): Treatment group 1 (300 mcg/kg/day) of a two-arm, dose-escalation pilot feasibility trial of TXA127 (Angiotensin 1-7) in subjects undergoing double cord blood transplantation for the treatment of a variety of hematologic malignancies for whom there is no available therapy with substantive anti-disease effect.
  Interventions: Drug: TXA127 300 mcg/kg/day
- TXA127 1000 mcg/kg/day (Experimental): Treatment group 2 (1000 mcg/kg/day) of a two-arm, dose-escalation pilot feasibility trial of TXA127 (Angiotensin 1-7) in subjects undergoing double cord blood transplantation for the treatment of a variety of hematologic malignancies for whom there is no available therapy with substantive anti-disease effect.
  Interventions: Drug: TXA127 1000 mcg/kg/day

INTERVENTIONS:
Drug: TXA127 300 mcg/kg/day — Injection, 300 mcg/kg/day for 28 days
  Arms: TXA127 300 mcg/kg/day
Drug: TXA127 1000 mcg/kg/day — Injection, 1000 mcg/kg/day for 28 days
  Arms: TXA127 1000 mcg/kg/day

SUMMARY:
The purpose of this study is to evaluate the effect of TXA127 on neutrophil and platelet counts in adult patients who have undergone a double cord blood transplant. The study will also evaluate the effect of TXA127 on chemotherapy-induced mucositis, an inflammation of the mucous membranes in the digestive tract (mouth to anus) and immune reconstitution which helps patients fight infections. For patients undergoing CBT, both neutrophil and platelet normalization and immune reconstitution can be delayed. TXA127 has shown to be well tolerated by patients and appears to induce a rapid production of neutrophils and platelets in the bloodstream as well as increase the immune system components. It has also been shown to reduce the severity of chemotherapy-induced mucositis.

DETAILED DESCRIPTION:
Cord blood as a hematopoietic stem cell source has multiple advantages. Cord blood is normally discarded at birth and can easily be collected and stored. Availability of numerous CB banks has resulted in genetically diverse CB units including those from non-Caucasians. Once a suitable CB unit is located, confirmatory typing can be quickly performed and a donor unit can be shipped to the transplant center. Furthermore, because a CB graft results in a lower incidence of graft-versus-host-disease, one or two antigen-mismatched units are acceptable for transplantation. Despite these advantages, CB has a significant drawback which is that the number of hematopoietic stem cells obtained from a unit of CB is significantly lower than from a bone marrow (BM) harvest or peripheral blood stem cell (PBSC) harvest. Both engraftment and immune reconstitution are delayed in patients undergoing CB transplant. TXA127 is pharmaceutically-formulated angiotensin 1-7, a non-hypertensive derivative of angiotensin II (which contains the 8th amino acid conferring receptor binding to blood pressure receptors). TXA127 has multilineage effects on hematopoietic progenitors in vitro and in vivo. The hematopoietic properties demonstrated in preclinical and clinical studies support the investigation of TXA127 to reduce time to neutrophil and platelet engraftment following transfusion of limited number of CD34+ cells.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Acute Myelogenous Leukemia (AML) past first remission, in first or subsequent relapse, induction failure, or in first remission with high-risk for relapse (with high-risk cytogenetics or presence of flt3 mutation or secondary leukemia from prior chemotherapy)
* Myelodysplastic Syndrome or Myelofibrosis of intermediate or high-risk
* Acute Lymphoblastic Leukemia (ALL): Induction failure, fist complete remission with Philadelphia chromosome or translocation (4:11), hypodiploidy and or evidence of minimal residual disease by flow cytometry, second or third complete remission or second relapse
* Chronic Myelocytic leukemia (CML): Second chronic phase or accelerated phase
* Non-Hodgkin's Lymphoma (NHL): Induction failures, second or third complete remission or relapse
* Hodgkin's Lymphoma (HL): Induction failures, second or third complete remission or relapse
* Chronic Lymphocytic leukemia (CLL): Progressive disease following standard therapy
* Other hematologic malignancies which meet investigational site standards for cord blood transplant
* Subjects must be at least 18 years of age
* Subjects must have ECOG status of ≤ 2
* Subjects with bone marrow blasts ≤ 10%
* Subjects must have adequate major organ function
* Male and Female Subjects capable of reproduction must agree to use contraceptive methods during the course of the study and for 2 months following the last administration of study drug
* Cord blood requirements: a) Unrelated CB will be used as a source of hematopoietic support if a 7/8 or 8/8 related or 8/8 unrelated bone marrow donor is not available, or if the tempo of the subject's disease dictates it is not in the subject's best interest to wait for an unrelated marrow donor to be procured. b) Subjects must have two CB units available which are matched with the subject at 4/6, 5/6, or 6/6 HLA class I (serological) and II (molecular) antigens. Each unit must contain at least 1 x 10^7 total nucleated cells/kg recipient body weight (pre-thaw).

Exclusion Criteria:

* Subjects who received antineoplastic treatment including chemotherapy, immunotherapy and radiation therapy ≤ 2 weeks prior to Screening Period
* Subjects who underwent prior total body irradiation
* Subjects who received prior allogeneic hematopoietic cell transplants
* Subjects seropositive for HIV, Hepatitis B or Hepatitis C
* Female subjects who are pregnant or breastfeeding
* Subjects who have received an investigational drug within 30 days of projected first administration of study drug (Day 0)
* Subjects with current alcohol use, illicit drug use, or any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the subject's ability to comply with the study requirements or visit schedule
* Subjects with known hypersensitivity to TXA127
* Subjects with uncontrolled medical or psychiatric condition which would limit informed consent
* Subjects with a willing and appropriate HLA-matched related marrow donor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Safety of TXA127 (Angiotensin 1-7) in subjects undergoing double cord blood transplantation | 100 days post-transplantation
  The safety and tolerability profile of TXA127 will be provided by descriptively summarizing, at a minimum, the following outcomes: 1) number and proportion of patients with adverse events presented by preferred term, by system organ class (SOC), and by severity grade and relationship to TXA127, as assessed by the Investigator; 2) number and proportion of patients terminating TXA127 due to adverse events related to TXA127; 3) Day 100 treatment-related mortality (TRM) rate; 4) Day 100 mortality rate; 5) number of red blood cell and other blood component transfusions; 6) incidence of infection.

SECONDARY OUTCOMES:
Platelet transfusion requirements | 100 days post-transplantation
  Platelet transfusion requirements based on units of platelets transfused and days of platelet transfusions
Immune reconstitution | 100 days post-transplantation
  Immune reconstitution will be assessed via the measurement of peripheral blood concentrations of CD3+, CD4+, CD8+, CD19+, and CD56+ cells (performed at Study Days 62 and 100).
Incidence, duration, and severity grade of mucositis | 100 days post-transplantation
  Incidence of mucositis is defined by the occurrence of least one adverse event with MedDRA preferred term that includes "mucositis" or "stomatitis". The severity grade will be determined by NCI-CTCAE.
Incidence, duration, and severity grade of acute graft-vs-host-disease (aGVHD) | 100 days post-transplantation
  Incidence, severity and duration of aGVHD will be reported as a proportion (with 95% CIs) of subjects with Grade II-IV aGVHD. All incidents of aGVHD will at a minimum be listed, with the severity and time course included.
Time to engraftment/recovery | 100 days post-transplantation
  Time to neutrophil engraftment and platelet recovery

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States